CLINICAL TRIAL: NCT07130981
Title: Evaluation of Body Composition, Psychosocial Factors, and Drug-Related Problems in Relation to Clinical Progression in Cancer Patients Receiving Immune Checkpoint Inhibitors
Brief Title: Body Composition and Psychosocial Factors in ICI-Treated Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, İzgi Bayraktar, PhD candidate, Hacettepe University
Other Study IDs: SBA 25/672
Record Dates: First submitted 2025-08-06; First posted 2025-08-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Psychosocial Functioning; Treatment Side Effects; Cachexia
MeSH Terms: conditions — Neoplasms; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Evaluation of the effects of body composition, psychosocial factors, and drug-related problems on clinical progression (such as toxicity, treatment response, and quality of life) in cancer patients treated with immune checkpoint inhibitors

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Having undergone a CT scan (at the L3 level) prior to treatment
* No severe mental disorder and able to communicate effectively
* Provided written informed consent

Exclusion Criteria:

* Did not provide written informed consent
* Patients deemed unsuitable by the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients initiating immune checkpoint inhibitor therapy (ipilimumab, nivolumab, pembrolizumab, atezolizumab, or avelumab) at the Medical Oncology Outpatient Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Body composition evaluation | Patient recruitment is planned to occur over a 6-month period. Each participant will be followed for a maximum duration of 6 months from the initiation of immunotherapy.
  Body Composition Parameters Description: Muscle area, muscle index, muscle density, lean body mass, and combined indices derived from routine abdominal imaging at the L3 vertebral level.
  Unit of measure: cm², cm²/m², Hounsfield units (HU), kilograms. Tool: Routine clinical imaging analysis.

SECONDARY OUTCOMES:
Cachexia and psychosocial factors evaluation | Throughout 6 months of follow-up.
  Cachexia Risk Scores Description: Composite scores reflecting cachexia status, based on multidimensional clinical and biochemical indicators.
  Unit of measure: Scoring system Tool: Validated cachexia scoring system. Psychosocial Factor Scores Description: Scores representing levels of depression, anxiety, stress, and distress, assessed through validated self-report questionnaires.
  Unit of measure: Questionnaire scores (scale ranges such as 0-21 or 0-10). Tool: Validated patient-reported outcome measures.
Drug Related Problems | Throughout 6 months of follow-up.
  Drug-Related Problems (DRPs) Description: Number and type of drug-related problems identified during treatment follow-up.
  Unit of measure: Count (number of problems per patient). Tool: Pharmaceutical Care Network Europe (PCNE) classification system. Immune-Related Adverse Events (irAEs) Description: Incidence and severity of immune-related adverse events occurring during immunotherapy.
  Unit of measure: Percentage of patients; severity graded 1-5. Tool: Common Terminology Criteria for Adverse Events (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Pharmacy, Department of Clinical Pharmacy, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No